CLINICAL TRIAL: NCT02366013
Title: A Phase 1 Clinical Trial of the Safety and Immunogenicity of an Oral, Replicating Adenovirus 26 Vector Vaccine for HIV-1 (rcAd26.MOS1.HIV-Env) in Healthy HIV-1-uninfected Adults
Brief Title: Trial of the Safety and Immunogenicity of an Oral, Replicating Ad26 Vectored HIV-1 Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: University of Rochester (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: rcAd001/IAVI R001
Record Dates: First submitted 2015-02-04; First posted 2015-02-19 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: HIV
Keywords: HIV; HIV Prevention; HIV Vaccine; Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental): 1 dose of rcAd26.MOS1.HIV-Env 1x10^8 vp or placebo
  Interventions: Biological: rcAd26.MOS1.HIV-Env 1x10^8 vp
- Group 2 (Experimental): 1 dose of rcAd26.MOS1.HIV-Env 1x10^9 vp or placebo
  Interventions: Biological: rcAd26.MOS1.HIV-Env 1x10^9 vp
- Group 3 (Experimental): 1 dose of rcAd26.MOS1.HIV-Env 1x10^10 vp or placebo
  Interventions: Biological: rcAd26.MOS1.HIV-Env 1x10^10 vp
- Group 4 (Experimental): 1 dose of rcAd26.MOS1.HIV-Env 1x10^11 vp or placebo
  Interventions: Biological: rcAd26.MOS1.HIV-Env 1x10^11 vp

INTERVENTIONS:
Biological: rcAd26.MOS1.HIV-Env 1x10^8 vp — 1 oral capsule, 1x10^8 vp/capsule or 1 placebo capsule; 5:1 vaccine:placebo
  Arms: Group 1
Biological: rcAd26.MOS1.HIV-Env 1x10^9 vp — 10 oral capsules, 1x10^8 vp/capsule or 10 placebo capsules; 5:1 vaccine:placebo
  Arms: Group 2
Biological: rcAd26.MOS1.HIV-Env 1x10^10 vp — 1 oral capsule, 1x10^10 vp/capsule or 1 placebo capsule; 5:1 vaccine:placebo
  Arms: Group 3
Biological: rcAd26.MOS1.HIV-Env 1x10^11 vp — 10 oral capsules, 1x10^10 vp/capsule or 10 placebo capsules; 5:1 vaccine:placebo
  Arms: Group 4

SUMMARY:
This is a dose escalation study to test the safety and immunogenicity of an oral HIV-1 vaccine.

DETAILED DESCRIPTION:
This study is a phase I dose-escalation randomized, double blind, placebo-controlled study designed to evaluate the safety and immunogenicity of rcAd26.MOS1.HIV-Env, an oral replicating adenovirus 26 vector vaccine in healthy HIV-1 uninfected adults. The vaccine will be administered orally at a single time point (Day 0) at one of four dose levels depending on study group: 1 x 10^8 virus particles (vp), 1 x 10^9 vp, 1 x 10^10 vp and 1 x 10^11 vp. Volunteers will be randomized to vaccine: placebo in a 5:1 ratio in each group.

Volunteers will be screened up to 56 days before vaccination and will be followed for 12 months after vaccination.

Because the vaccine is replication competent, volunteers will be housed in an isolation unit from day -2 through day 9. Household contacts will also be enrolled and tested for possible transmission.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years old.
* Ability and willingness to provide informed consent.
* Complete an assessment of understanding
* Available for the duration of the trial, including willingness to be kept in an isolation facility
* From Day 10 through 4 months following vaccination must reside alone or with no more than 2 adults (age 18-60) and no minors under age 18
* Good general health as shown by medical history, physical exam, and screening
* Willing to undergo HIV testing and willing to receive risk reduction counseling
* All female volunteers must be willing to undergo urine pregnancy tests
* Sexually active males must be willing to use an effective method of contraception until at least 4 months after vaccination
* Women of child bearing potential commit to use an effective method of contraception when sexually active with males for 4 months after vaccination
* Willing to forgo donations of blood or any other tissues during the study and, for those who test HIV positive due to trial vaccination (vaccine-induced HIV seroreactivity), until the anti-HIV antibody titers become undetectable
* Low risk for HIV infection and willing to maintain low-risk behavior for the trial duration

Exclusion Criteria:

* Confirmed HIV-1 or HIV-2 infection; confirmed HCV, HBV, or syphilis infection
* Current or planned participation in another clinical trial of an experimental agent during the study period
* Pregnant or lactating
* Significant acute or chronic disease, including inflammatory bowel disease or other chronic gastrointestinal disease, immunodeficiency syndrome, or condition requiring immunosuppressant medications
* Use of anticancer, antituberculosis or other medications considered significant by the investigator within the previous 6 months
* Receipt of live-attenuated vaccine within the previous 60 days or planned receipt within 60 days after vaccination with Investigational Product (within 14 days for live attenuated influenza vaccine [LAIV]); or receipt of other vaccine (e.g., influenza, pneumococcal), allergy treatment with antigen injections or tuberculin skin test within the previous 14 days or planned receipt within 14 days after vaccination with Investigational Product
* Receipt of blood transfusion or blood-derived products within the previous 3 months
* Receipt of HIV vaccine(s) in a prior HIV vaccine trial.
* Previous severe local or systemic reactions to vaccination
* History of splenectomy
* History of seizure in the last 3 years
* Known autoimmune disease
* Asthma other than mild, well-controlled asthma.
* Diabetes mellitus type 1 or type 2
* Thyroidectomy, or thyroid disease requiring medication during the last 12 months
* Angioedema within the last 3 years if episodes are considered serious or have required medication within the last 2 years
* Hypertension
* Body mass index (BMI) ≥ 40
* Bleeding disorder diagnosed by a doctor
* Malignancy (Not excluded: a volunteer with a surgical excision and subsequent observation period that in the investigator's estimation has a reasonable assurance of sustained cure or is unlikely to recur during the study period)
* Psychiatric condition that compromises safety of the volunteer or precludes compliance with the protocol
* All healthcare workers with direct patient contact
* Childcare worker who has direct contact with children
* Individuals employed as food handlers or otherwise engaged in the preparation or delivery of food outside of their place of residence
* Positive urine toxicology test

Household contacts 18-60 years of age are also evaluated for eligibility with a more abbreviated list of inclusion/exclusion criteria.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as measured by number of volunteers reporting the following: | 4 Months post-vaccination
  * Any adverse events within 4 months following vaccination (SAEs within 12 months following vaccination)
  * Moderate or greater unsolicited adverse events related to study product (i.e., suspected adverse reactions) within 4 weeks post-vaccination
  * Moderate or greater solicited reactions within 9 days post-vaccination

SECONDARY OUTCOMES:
Proportion (95%CI) of volunteers per dose group with positive shedding responses and mean response per group with 95% CI. | 28 days
  o Rectal/oral shedding: real-time PCR for rcAd26.MOS1.HIV-Env at 1, 2, 3, 4, 5, 6, 7, 8, 9, 12, 17, 21, 7, 12, 21, and 28 days after vaccination.
Proportion of volunteers per dose group with positive immunological responses and mean response (e.g. GMT) per group with 95% CI. | 12 Months
  * Cellular immunogenicity: Env-specific ELISPOT responses at 4 weeks after vaccination.
  * Humoral immunogenicity: Env-specific binding antibody titers at 4 weeks after vaccination.
  * Durability of responses: immunogenicity assays at 4, 8 and 12 months after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: John Treanor, MD, Principal Investigator — University of Rochester; Kathryn Stephenson, MD, MPH, Study Chair — Beth Israel Deaconess Medical Center
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Derived] Stephenson KE, Keefer MC, Bunce CA, Frances D, Abbink P, Maxfield LF, Neubauer GH, Nkolola J, Peter L, Lane C, Park H, Verlinde C, Lombardo A, Yallop C, Havenga M, Fast P, Treanor J, Barouch DH. First-in-human randomized controlled trial of an oral, replicating adenovirus 26 vector vaccine for HIV-1. PLoS One. 2018 Nov 14;13(11):e0205139. doi: 10.1371/journal.pone.0205139. eCollection 2018. PMID 30427829